CLINICAL TRIAL: NCT06857279
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-HNSCC201
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma of Head and/or Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HLX43 DOSE 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 1
- HLX43 DOSE 2 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 2
- HLX43 DOSE 3 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 3

INTERVENTIONS:
Drug: HLX43 DOSE 1 — Dose 1; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 1
Drug: HLX43 DOSE 2 — Dose 2; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 2
Drug: HLX43 DOSE 3 — Dose 3; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 3

SUMMARY:
The study is being conducted to to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC). In this study, eligible subjects will be randomized at 1:1:1 ratio, and the patients will be administered with HLX43 at different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements;
2. Aged ≥ 18 years and ≤ 75 years at the time of signing the ICF, male or female;
3. Patients with histologically confirmed recurrent/metastatic head and neck squamous cell carcinoma who have failed previous systemic treatment;
4. At least one measurable lesion as per RECIST 1.1 within 4 weeks prior to randomization;
5. Subjects who agree to provide archived tumor tissue specimens that meets the testing requirements or agree to undergo a biopsy;
6. The following conditions must be met in terms of the time of the first administration of the investigational product: at least 3 weeks (or 5 half-lives of the drug, whichever is shorter) from the previous major surgery, medical device treatment, locoregional radiotherapy (except for palliative radiotherapy for bone lesions), cytotoxic chemotherapy, immunotherapy, or biological product therapy; at least 2 weeks from the previous hormone therapy or small molecular targeted therapy; at least 1 week from the administration of the traditional Chinese medicine for anti-cancer indications or minor surgery; and recovery of treatment-induced AEs to Grade ≤ 1;
7. ECOG PS score of 0-1 within 1 week prior to randomization;
8. Life expectancy > 3 months;
9. Adequate organ functions as confirmed by laboratory tests within 1 week prior to randomization;
10. Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last dose of the investigational product; female subjects of childbearing age must be negative for pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

Patients who meet any of the following criteria are not allowed to be enrolled:

1. Patients with head and neck tumor who are indicated for locoregional radical treatment;
2. Patients with primary nasopharyngeal carcinoma;
3. Imaging examination shows that the tumor has invaded or surrounded the large blood vessels of the chest, neck, and pharynx, and there is imaging evidence that entering the study will induce risks of hemorrhage;
4. History of any second malignancy within 2 years prior to randomization, ;
5. Occurrence of Grade ≥ 3 immune-related adverse events (irAEs) during prior immunotherapy;
6. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
7. Patients who have newly diagnosed or clinically symptomatic brain metastases, spinal cord compression, or cancerous meningitis, or uncontrolled brain or spinal cord metastases that have been evidenced;
8. Patients with previous or current interstitial pneumonia, pneumoconiosis, drug-related pneumonitis, or severe lung function impairment that may interfere with the detection and management of suspected drug-related pulmonary toxicity; patients with radiation pneumonitis within 6 months;
9. Patients with any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months (except lacunar infarction, slight cerebral ischemia, or transient ischemic attack); (4) poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia's formula); (5) poorly-controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg after active treatment);
10. Patients with active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to randomization;
11. Patients who have used potent CYP2D6 or CYP3A inhibitors or inducers within 2 weeks prior to randomization;
12. Patients who have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 2 weeks prior to randomization;
13. Patients with known active or suspected autoimmune diseases;
14. Patients who have received live vaccine or live attenuated vaccine within 4 weeks prior to randomization;
15. Patients who are known to have severe anaphylaxis to macromolecular protein preparations/monoclonal antibodies or are allergic to any component in the formulation of the investigational product;
16. Patients with active tuberculosis;
17. Patients with a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or history of organ transplantation;
18. Patients with active HBV or HCV infection or HBV/HCV co-infection;
19. Pregnant or lactating women;
20. Patients who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by INV according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by the IRRC according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC according to the RECIST v1.1 criteria.
OS | From randomization to death from any cause (up to approximately 36 months)
  Overall Survival
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0, vital signs and clinical laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, Dr, Principal Investigator — Fudan University; Man Hu, Dr, Principal Investigator — Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences
Locations (2):
- China (2):
  - Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai